CLINICAL TRIAL: NCT05229172
Title: Prospective Multicenter Observational Study of the Safety and Performance of Fabian Ventilator System Volume Guarantee Mode in Routine Use
Brief Title: Fabian Prospective Assessment of Volume Guarantee (Fabian PaVoG)
Acronym: PaVoG
Status: Completed | Type: Observational
Sponsor: Vyaire Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-21-003-PaVoG
Record Dates: First submitted 2021-11-22; First posted 2022-02-08 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2022-01

CONDITIONS: Respiratory Insufficiency in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Volume Targeted Ventilation — There is no study specific intervention planned. Procedures will be conducted according to standard of care of each participating hospital and the instructions for use of the study device.

SUMMARY:
This study is planned as a part of the post market clinical follow-up (PMCF) on a CE marked product and will provide performance data on the Volume Guarantee function of the fabian ventilator in daily clinical routine.

DETAILED DESCRIPTION:
PaVoG study is a prospective, multicenter, single-cohort post market observational study.

The study procedures will be conducted according to standard of care of each participating hospital and the instructions for use of the study device.

To allow data collection, an Informed Consent Form will be obtained from each study participant/ legally authorized representative, if required by the local Ethical Committee. Ventilator data will be recorded in the hospital's data capture system or on a study laptop provided by the Sponsor.

Each patient will be clinically evaluated according to hospital standard of care. If inclusion and exclusion criteria are met, and the investigative team is available the patient will be enrolled.

Study duration for an individual patient will differ, depending on the time spent on fabian ventilator with Volume Guarantee mode on.

It is anticipated that for most will be between 2-4 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient ventilated with fabian ventilator (conventional or HFOV) with VG mode active.
* The anticipated use of VG mode is at least 12 hours
* Informed Consent given by parents or guardians according to the process approved by the local research ethical committee

Exclusion Criteria:

* Patients with severe airflow obstruction and intracranial hypertension
* Decision documented to give palliative neonatal care.
* The clinical care team does not agree with inclusion of the infant to the study

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Infants in the intensive care unit setup receiving respiratory support from fabian ventilator with Volume Guarantee (VG) mode active.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
In Conventional Mechanical Ventilation (CMV) with Volume Guarantee (VG) - Relationship between tidal volume set vs tidal volume observed (Volume guarantee mode) | through study completion, an average of 2 - 4 days
  Difference between set and observed expired tidal volume (VTe), average - on the patient level and breath-to-breath variability will be reported
In High Frequency Oscillatory Ventilation with Volume Guarantee (HFOV-VG)- Relationship between the set and observed tidal volume of oscillations (VThf) during HFOV-VG | through study completion, an average of 2 - 4 days
  Difference between the set and observed VThf (average and variability)

SECONDARY OUTCOMES:
Ventilator Performance - Relationship between the set and observed Positive End-Expiratory Pressure (PEEP) and Continuous Positive Airway Pressure (CPAP) | through study completion, an average of 2 - 4 days
  Difference between set and observed PEEP (average and variability)
Ventilator Performance - Variability of Peak Inspiratory Pressure (PIP) during Volume Guarantee (VG) ventilation | through study completion, an average of 2 - 4 days
  Standard deviation of PIP will be reported
Ventilator Performance - Relationship of Peak Inspiratory Pressure (PIP) during Volume Guarantee (VG) ventilation to the set maximum allowed inflating pressure (Pmax) | through study completion, an average of 2 - 4 days
  Mean difference between Pmax and PIP will bereported
Ventilator Performance - Relationship between the set and observed mean airway pressure (MAP) during HFOV | through study completion, an average of 2 - 4 days
  Difference between the set and observed MAP (average and variability)
Ventilator Performance - Relationship between the set and observed Fraction of Inspired Oxygen (FiO2) | through study completion, an average of 2 - 4 days
  Difference between the set and observed FiO2 (average and variability)
Ventilator Performance - Reason(s) to switch off Volume Guarantee | through study completion, an average of 2 - 4 days
  The reason for stopping Volume Guarantee will be documented in the case report form
Ventilator Safety - Device failure rate | through study completion, an average of 2 - 4 days
  Malfunction of the investigational device necessitating removal of a neonate to another ventilation mode or ventilator
Ventilator Safety - Descriptive statistical analysis of all ventilator alarm events | through study completion, an average of 2 - 4 days
  A summary table presenting number, type and duration of ventilator alarms within study population
Ventilator Safety - Number of study participants with device related adverse events | through study completion, an average of 2 - 4 days
  Number of malfunction of the investigational device leading to potential or actual patient harm
Exploratory analysis - Relationship between end-tidal CO2 (etCO2) or transcutaneous CO2 (tcCO2) and Partial Pressure of Carbon Dioxide (pCO2) in blood gases (capillary and arterial) in infants of different clinical characteristics | through study completion, an average of 2 - 4 days
  Correlation between average end-tidal CO2 (etCO2)/ transcutaneous CO2 (tcCO2) and blood gas Partial Pressure of Carbon Dioxide (pCO2); Bland-Altman plots
Exploratory analysis - Relationship between expired tidal volume (VTe) or Minute Volume (MV) and end-tidal CO2 (etCO2) or Partial Pressure of Carbon Dioxide (pCO2) or transcutaneous CO2 (tcCO2) in infants of different clinical characteristics | through study completion, an average of 2 - 4 days
  Correlation analysis between expired tidal volume and CO2 measurements per patient
Exploratory analysis - Feasibility of volumetric capnography | through study completion, an average of 2 - 4 days
  A summary table presenting duration, accuracy and availability of volumetric capnography data in neonatal patients
Analysis of patient-ventilator interactions - Analysis of number of triggered and backup ventilator inflations per patient | through study completion, an average of 2 - 4 days
  The impact of set ventilator rate and expiratory time on the number of triggered and backup inflations.
Analysis of patient-ventilator interactions - analysis of Tidal Volume of triggered and back inflations | through study completion, an average of 2 - 4 days
  Tidal volume of triggered and backup ventilator inflations will be analyzed and compared
Analysis of patient-ventilator interactions - Contribution of the infant to the total minute ventilation via spontaneous breathing between ventilator inflations per patient | through study completion, an average of 2 - 4 days
  The impact of ventilator modes and settings will be analyzed and compared
Analysis of patient-ventilator interactions - Ventilator-patient asynchronies per patient | through study completion, an average of 2 - 4 days
  The occurrence and frequency of inspiratory hold during time cycled ventilation. The frequency of interrupted expirations. Occurrence and frequency of incomplete expiration during neonatal ventilation. Calculation of asynchrony index per patient and for study population.

CONTACTS AND LOCATIONS:
Overall Officials: Gusztav Belteki, MD, PhD, Study Chair — Cambridge University Hospitals NHS Trust
Locations (5):
- University Medical Center Amsterdam, The Netherlands, Amsterdam, Netherlands
- Poland (3):
  - Szpital Położniczo - Ginekologiczny Ujastek, Krakow
  - Ginekologiczno-Położniczy Szpital Kliniczny Uniwersytetu Medycznego im. Karola Marcinkowskiego, Poznan
  - Centre of Postgraduate Medical Education, SPSK im prof.W.Orłowskiego, Warsaw
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No